CLINICAL TRIAL: NCT01446055
Title: Transplantation of Autologous BM-MNC Processed by ResQ Separator and Conventional Manual Method for Patients With Chronic Limb Ischemia: a Multi-center Randomized Controlled Trial
Brief Title: Safety and Efficacy Study of Autologous BM-MNC Processed by Two Methods for Treating Patients With Chronic Limb Ischemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Thermogenesis Corp. (Industry); Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yong-Quan Gu, Director of Vascular Surgery Department, Principal Investigator, Clinical Professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TGResQ082011
Record Dates: First submitted 2011-09-23; First posted 2011-10-04 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease; Buerger's Disease
Keywords: Peripheral arterial disease; Buerger's disease; atherosclerotic arterial occlusion; bone marrow mononuclear cell; chronic limb ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Thromboangiitis Obliterans

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ResQ process group (Experimental): Autologous BM-MNC is enriched with ResQ process(an automatic cell separator). Then the cell product is transplanted into the ischemia limbs of a patient.
  Interventions: Device: ResQ processed bone marrow sample
- Ficoll-based conventional method (Active Comparator): A conventional method based on Ficoll cell separation is used to process bone marrow.
  Interventions: Device: Ficoll conventional cell processing method

INTERVENTIONS:
Device: ResQ processed bone marrow sample — Autologous bone marrow is processed with ResQ at point of care, prior to the transplantation
  Arms: ResQ process group
Device: Ficoll conventional cell processing method — Comparison of different cell processing methods
  Arms: Ficoll-based conventional method

SUMMARY:
Using autologous bone marrow mononuclear cells (BM-MNC) to treat patients with chronic limb ischemia has been proved safe and effective. However, processing bone marrow by Ficoll density gradient centrifugation is not only time consuming but also expensive. Manually processing of bone marrow also results in large variation in therapeutic cell quantity and quality which directly leads deviation of safety and efficacy of the cell therapy. This study is aiming to compare an automated bone marrow processing system with a conventional manual method in term of safety and efficacy.

DETAILED DESCRIPTION:
Using autologous bone marrow mononuclear cells (BM-MNC) to treat patients with chronic limb ischemia has been proved safe and effective. However, processing bone marrow by Ficoll density gradient centrifugation is not only time consuming but also expensive. Manually processing of bone marrow also results in large variation in therapeutic cell quantity and quality which directly lead deviation of safety and efficacy of the cell therapy. This study is aiming to compare an automated bone marrow processing system with a conventional manual method in term of safety and efficacy.

ResQ system developed by Thermogenesis in USA provides an automatic cell processing system for bone marrow. The system takes less than 30 minutes to concentrate the therapeutic mononuclear cells including stem cells in a closed system without adding any additive such as separation reagent (Ficoll). The system also be able to be operated at point of care.

The study is designed to prove no inferior of safety and efficacy of bone marrow cells processed by ResQ to those of cells using conventional manual method. The conventional manual method is involved Ficoll density gradient centrifugation and cell washing stems in an open system. Each of test arms (ResQ vs manual method) consists of 25 patients. The primary outcome is safety which is measured by cell treatment-related adverse events. The secondary endpoints include resting ankle-brachial pressure index (ABI)and toe brachial pressure index (TBI) , transcutaneous oxygen pressure (TcPO2), claudication distance, rest pain scale evaluation, collateral vessel scale, etc.

ELIGIBILITY:
Inclusion Criteria:

1. fontaine's stage 2-4 or resting ABI <0.7
2. age between 20 and 80 years old
3. sign informed consent, voluntary subjects
4. diagnosis of lower extremity arterial occlusive disease, or diabetic lower limb ischemia, or Buerger's disease

Exclusion Criteria:

1. poorly controlled diabetes (HBA1c> 7.0%) and proliferative retinopathy (III-IV stage)
2. malignancy history in the past five years or serum level of tumor markers elevated more than doubled
3. severe heart, liver, kidney, respiratory failure or poor general condition can not tolerate BM-MNC transplantation
4. serious infections (such as cellulitis, osteomyelitis, etc.)or gangrene that a major amputation cannot be avoided
5. aortic or iliac or common femoral artery occlusion
6. pregnant female, or reproductive age female who wants to give birth throughout the course of the study
7. life expectancy less than a year

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Cell treatment-related adverse event | 2-wk after bone marrow transplantation
  1. Temperature,Pulse,Respiration,Blood Pressure
  2. Routine analysis of blood and urine,
  3. Liver function(ALT：alanine aminotransferase,AST：aspartate transferase), Renal function(Blood urea nitrogen,Creatinine;) Function of coagulation(APTT,PT,Fib,TT）
  4. ECG（Electrocardiography）
  5. local inflammatory response
  6. Cell-treatment related death
  7. Cell-treatment related unexpected amputation.

SECONDARY OUTCOMES:
ulcer size | Post bone marrow transplantation: 1, 3, 6, 12 months
  Measuring ulcer area (cm2) and depth (mm)of limb :
  For each ulcer , photographically record the area and depth with a ruler in order to calculate the ulcer area in square millimeters.
rest pain score. | Post bone marrow transplantation: 1，3, 6, 12 months
  Scoring the rest pain based on the degree of pain as following five scales):
  0 level-0 point: no pain;
  1. level-1 point: occasional pain which can be recalled;
  2. level-2 points: the pain often but can be tolerated, without or with a little analgesics;
  3. level-3 points: often with need of general analgesics;
  4. level -4 points: affect sleeping due to the pain, general pain medication being difficult to alleviate.
  Before transplantation: points; after transplantation: points.
cold sensation score | Post bone marrow transplantation:,1，3, 6, 12 months
  based on a sense of cold as following five scales: 0 level-0 point: no cold sensation;
  1. level-1 point, or : Accasionally cold feeling;
  2. level-2 points: Often with cold feeling;
  3. level-3 points: significantly cold feeling. and can be significantly improved when using a local insulation.
  4. level-4 points: significantly cold feeling，and can not be significantly improved when using a local insulation.
claudication distance (m) | Post bone marrow transplantation:1, 3, 6, 12 months
  Measurement of claudication distance (m)： For patients with intermittent claudication, treadmill exercise test (no tilt, speed 3km/hr) is employed to measure claudication distance.
Resting ABI | Post bone marrow transplantation: 1,3, 6, 12 months
  Measurement of ABI(ankle brachial index, ABI):
  Measure arterial pressure with a laser Doppler, and then calculate the ankle-brachial index, that is a ratio of ankle arterial blood pressure to brachial arterial blood pressure at rest.
Resting TcPO2 (mmHg) | Post bone marrow transplantation:1, 3, 6, 12 months
  Transcutaneous oxygen pressure(TcPO2) should be measured at the same site in the ischemic limb at rest.
Collateral vessel score | Post bone marrow transplantation: 1,3, 6, 12 months
  Collateral vessel score:
  Using DSA(Digital subtraction angiography)or CTA(computed tomographic angiography) to score the collateral vessel formation.
  A mean score is obtained for each ischemic limb by 3 independent interventionists based on the following 4 level score:
  0 (no new collateral vessels)
  * 1 (A little new collateral vessels)
  * 2 (moderate new collateral blood vessels)
  * 3 (Rich new collateral vessels)
Amputation rate | Post bone marrow transplantation:1, 3, 6, 12 months
  Amputation rate and level is recorded.
Skin microcirculation measurement | 1,3,6,12 months post transplantation
  using PeriMed "laser-Doppler flowmetry" measure the skin microcirculation on the same site in the ischemic limb at rest.
Resting TBI | Post bone marrow transplantation: 1,3, 6, 12 months
  Measurement of TBI（Toe Brachial Index):
  Measure arterial pressure with a laser Doppler, and then calculate Toe Brachial Index, that is a ratio of toe arterial blood pressure to brachial arterial blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Quan Gu, Dr., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuan Wu Hospital, Beijing, Beijing Municipality, China